CLINICAL TRIAL: NCT07010198
Title: Head-to-Head Comparison of Hepatocellular Cancer (HCC) Screening Strategies: A Prospective Population-Based Cohort Study in Zhongshan City
Status: Recruiting | Type: Observational
Sponsor: Zhongshan People's Hospital, Guangdong, China (Other)
Responsible Party: Principal Investigator, Mingfang Ji, Clinical Professor, Zhongshan People's Hospital, Guangdong, China
Other Study IDs: HCC-2025-01
Record Dates: First submitted 2025-05-20; First posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-05

CONDITIONS: Hepatocellular Cancer (HCC)
Keywords: Screening; Hepatocellular Cancer; aMAP
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- HCC Screening Dynamic Cohort: Local household-registered residents aged 35-64 years who are HBsAg-positive and have not been diagnosed with HCC prior to enrollment, residing in the study site communities of Zhongshan City
  Interventions: Diagnostic Test: Quantitative HBeAg Testing; Biological: Measurement Indicators Required for Risk Scoring in HCC Screening Strategies; Biological: Follow-Up Monitoring Parameters

INTERVENTIONS:
Diagnostic Test: Quantitative HBeAg Testing — Quantitative HBeAg Testing in Population-Based Primary Screening
Biological: Measurement Indicators Required for Risk Scoring in HCC Screening Strategies — REACH-B: Age, Sex, HBeAg status, ALT levels, and HBV DNA load; AGED: Age, Sex, HBeAg status, HBV DNA load; aMAP: Age, Sex, Albumin, Total Bilirubin, Platelet Count; aMAP 3.0: Age, Sex, Albumin, Total Bilirubin, Platelet Count, AFP and PIVKA-II.
Biological: Follow-Up Monitoring Parameters — AFP, Liver Ultrasound

SUMMARY:
Based on the preliminary retrospective validation of the efficacy of five HCC screening strategies(including conventional AFP combined with ultrasound-based general screening strategy, REACH-B, AGED, aMAPand aMAP 3.0 risk score) in Xiaolan Town, a head-to-head comparison for HCC screening is conducted in Zhongshan City, Guangdong Province. The study is a prospective, single-center, head-to-head trial aiming to enroll 4,500 HBsAg-positive individuals. It adopts a two-phase design of "HBV screening first, followed by HCC surveillance":Phase I: Recruitment of age-eligible populations at study sites for HBsAg screening to establish a high-risk cohort positive for hepatitis B surface antigen.Phase II: Implementation of uniform HCC surveillance (AFP combined with liver ultrasound every six months) for HBsAg-positive individuals, with concurrent application of different risk stratification models to evaluate risk levels and screening efficacy for each participant during follow-up.Furthurmore, based on baseline biological information and follow-up data, the study also aims to explore the development of a more effective risk prediction model for HCC.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily sign the informed consent form.
* Household registration in Zhongshan City, Guangdong Province.
* Aged 35 and above.
* Positive screening result for Hepatitis B surface antigen (HBsAg).

Exclusion Criteria:

* Previous history of liver cancer or liver transplantation.
* Pregnant women.
* Severe comorbidities (e.g., end-stage cardiopulmonary diseases, advanced malignancies).
* Individuals lacking legal capacity or unable to provide informed consent.

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Local household-registered residents aged ≥35 years, HBsAg-positive, with no prior diagnosis of HCC, residing in Zhongshan City.
Sampling Method: Non-Probability Sample
Enrollment: 4500 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of HCC | 3 years
  The number of newly diagnosed HCC cases divided by total person-years at risk during follow-up for each screening strategy.
Predictive performance (Sensitivity, Specificity, Positive Predictive value, AUC, etc.) | 3 years
  Sensitivity, specificity, positive predictive value(PPV) and area under the ROC curve (AUC) will be calculated to evaluate the discrimination of each model.
Risk stratification accuracy | 3 years
  Participants will be categorized into different risk strata (high, intermediate, low) by each model, and their observed HCC incidence will be compared to assess stratification accuracy.

SECONDARY OUTCOMES:
Screening positivity and referral rate | 3 years
  Proportion of participants identified as medium/high-risk and referred for further diagnostic imaging (e.g.,pathology/CT/MRI).
Stage distribution of HCC cases identified by different screening strategies | 3 years
Early detection rate of HCC cases identified by different screening strategies | 3 years
Number Needed to Screen (NNS) | 3 years
  Number of individuals needed to be screened to prevent one case of HCC.
Incremental Cost-Effectiveness Ratio (ICER) | 3 years
  The additional cost required to gain one extra QALY or to prevent one HCC case using a given model, compared with baseline strategy.
Time-dependent AUC or C-index | 3 years
  Model discrimination assessed at different time points using time-dependent ROC curves and concordance index (C-index).
Model performance in subgroups | 3 years
  Subgroup analyses to compare predictive performance of each model in different populations (e.g., by sex, age, ALT level, HBV DNA level).
Overall survival (OS) | 3 years
  Indicates whether the participant was alive at the end of follow-up and their survival duration.
Screening adherence | 3 years
  The proportion of participants who completed biannual AFP and ultrasound screenings as scheduled during follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan People's Hospital, Zhongshan, Guangdong, China